CLINICAL TRIAL: NCT03014154
Title: Effects of Video Training With Active Gambling Associated With Resistance Exercise Inflammatory and Functional Outcomes in Children Clinical Teaching Blind Randomized
Brief Title: Assessment of the Effects of Strenght Exercise With Active Video Game Games in Asthmatic Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Juliana Fernandes Barreto de Mendonça, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 907236/2014
Record Dates: First submitted 2015-10-13; First posted 2017-01-09 (Estimated); Last update posted 2017-12-05 (Actual); Status verified 2017-12

CONDITIONS: Pulmonary Diseases, Obstructive; Asthma
Keywords: video games; asthma; physical exercise
MeSH Terms: conditions — Lung Diseases, Obstructive; Asthma; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Video training Game (Active Comparator): Patients were submitted prior to the treadmill warming the 2kmh during 1° minutes before each session. Then held 30 minutes of aerobic interval training with video game (10 rounds of 3 minutes with 30 seconds of rest between each), followed by 5 minutes of cool-down again on the mat. The game used for training was the "reflex Ridge" Kinect Adventure (Xbox-360). At a higher level, it is necessary for the child to perform a greater number of jumps, squats, lateral movements and arm movements. All the activity was monitored against FC and SpO2. To determine the intensity of physical activity energy expenditure assessments were made. In which four are for the pre and post intervention evaluation and sixteen training sessions.
  Interventions: Other: Training
- Endurance muscle training (Active Comparator): Patients were submitted prior to the treadmill warming the 2kmh during 1° minutes before each session. Then held 30 minutes of aerobic interval training with video game (10 rounds of 3 minutes with 30 seconds of rest between each) followed by 5 minutes of cool-down again on the mat.Then the children were subjected to low intensity to endurance muscle training with 3 sets of 15 repetitions to upper limbs diagonally primitive and flexion and extension to lower lumbs. All the activity was monitored against FC and SpO2.To determine the intensity of physical activity energy expenditure assessments were made. In which four are for the pre and post intervention evaluation and sixteen training sessions.
  Interventions: Other: Training

INTERVENTIONS:
Other: Training

SUMMARY:
Asthma is a chronic inflammatory disease of the Airways of recurring character. The obstruction to the airflow carries the short-and long-term consequences that require prophylactic interventions and in emergency many times. The children due to immaturity of the respiratory system associated with the use of steroids suffer structural consequences, as for example, the physical deconditioning that intensifies the symptoms of the disease and affects negatively on the quality of life. Therefore, to set up a physical training program suitable for the paediatric population, using resources to increase adherence to the regular practice of exercises, can be the difference for the reduction of the number of exacerbations, the sensation of Dyspnea and the doses of medication, positively impacting the clinical picture of child asthmatic. The investigators conducted a randomized, blinded in order to evaluate the effects of training with active video game associated with resisted exercise the exercise in inflammatory and functional outcomes resisted in asthmatic children.

DETAILED DESCRIPTION:
OBJECTIVES:

General Objective:

o analyze the effects of a pulmonary rehabilitation program with aerobic exercise involving a VGA (Xbox 360) system associated with the exercise of strength and resistance to upper and lower limbs in patients susceptible to asthma.

Specific Objectives:

To evaluate the clinical control of asthma, quality of life, airway inflammation, exercise tolerance and energy expenditure in an aerobic training with videogame (Xbox 360) associated with strength training and resistance of upper and lower limbs .

Compare between training groups the results obtained through the evaluated variables.

MATERIAL AND METHODS:

Ethical and legal aspects:

This Protocol was approved by the Committee of Ethics in Research with Human Beings of the University Nove de Julho (Brazil), under the paragraph of opinion. 9072362014.

The rights must sign a Free and Informed Consent Term (TFCC) and all beings authorized to be removed at any time without any encumbrance. All study procedures are confidential.

Characterization of the study:

This is a clinical trial developed at the Laboratory of Functional Respiratory Analysis (LARESP) of Master and Post-Graduation in Rehabilitation Sciences of the University of Nove de Julho (UNINOVE).

Subject and Recruitment:

Patients will be recruited consecutively and selected for eligibility according to the proposed protocol, invited to the Hospital Set de Mandaqui (São Paulo, Brazil) and referred to LARESP (São Paulo, Brazil).

After consent for participation in the study through FICS signature, the patients will be submitted to evaluation. Assessments will be divided and two steps taken during the first week and training protocols commenced the following week.

Before and after the training protocols, the patients will be submitted to anthropometric and electrical bioelectrical impedance tests, will respond to quality of life questionnaires (PAQLQ) and clinical control of asthma, pulmonary function test, spirometry, respiratory muscle strength ), Fraction of Nitric Oxide Test (FeNO), incremental test for upper and lower limbs, through the 1 repetition maximal test (1RM) and functional capacity test by means of the treadmill test (Bruce protocol).

Reviews:

After consent for participation in the study, patients will be evaluated. Evaluations will be divided into two stages and will be conducted during the first week and training protocols will begin the following week.

After 8 weeks, patients will be submitted to the same initial evaluations.

Anthropometric:

Body weight will be obtained by digital scale (Filizola ®, Brazil). The height will be evaluated by a wall-mounted stadiometer (Wiso), with a resolution in millimeters. To obtain the Z score, we used the Anthro plus program, which uses World Health Organization (WHO) standards for Z score. BMI Z scores were used to classify obese or eutrophic children.

Body Composition:

The participants' body composition will be evaluated using a four-way electric bioimpedance scale, the mechanism currently supported as the most accurate for this. Biodynamic ™ Model 310 (Biodynamics Corporation Seattle WA, USA).

For the measurement of body composition foam placed four electrodes on patients' skin, previously cleaned with alcohol. Two electrodes were placed in the upper right corner (next to the digital metacarpophalangeal of the dorsal surface of the hand and another between the prominences of the distal radius and ulna) and another at the lower extremity also half of the body (a distal distal) Second between the medial and lateral malleolus of the ankle).

To perform the desired patient was instructed not to drink caffeinated beverages at least 12:00 before the test; Do not eat or drink in a period of 4:00 before the test, urinate 30 minutes before the test and do not perform physical activity 6:00 before the test.

Quality of life questionnaire:

The Pediatric Asthma Quality of Life Questionnaire (PAQLQ) is a health-related quality of life. It is the most used instrument for childhood asthma, being the questionnaire best known and validated for the Brazilian population and can be used in children and adolescents from 7 to 17 years. The PAQLQ consists of 23 questions divided into three areas, namely: physical activity limitation (five issues); Symptoms (10 questions) and emotions (eight questions). Responses were measured using a 7-point scale, where 1 indicates the maximum loss and 7 the loss.

Asthma Control Questionnaire:

The Asthma Control Questionnaire (ACQ) is a questionnaire to assess clinical control in asthmatic patients and consists of 7 questions, 5 related to asthma symptoms, the use of short-acting ß2 agonist as rescue medication and pre-bronchodilator Percentage Of FEV1 predicted. The ACQ score is the mean of these items and ranges from 0 (fully controlled) to 6 (out of control), obtained over a period of 7 days. The cutoff point for uncontrolled asthma is 2 points. The patient will be classified according to ACQ scores in controlled asthma (0.75), partially controlled (0.75 -1.5) and uncontrolled (1.5). A minimum clinical difference difference of 0.5 on a 7-point scale. The version used will be that of ACQ6.

Pulmonary function test:

The lung function test was performed through spirometry, which will analyze lung volumes, capacities and flows. The test consists of inspiratory and expiratory maneuvers performed using an Easy One ® brand spirometer, the previously calibrated NDD. For the test, three reproducible maneuvers will be obtained, according to the ATS recommendations. All tests will be conducted in an air-conditioned environment and the reference values used were those of Polgar, suitable for children, for classification purposes, as well as post-intervention evolution.

Respiratory muscular endurance (FMR):

The FMR will be evaluated by means of the manovacuometry, obtaining the maximum respiratory pressure (MIP and MEP), using an analog manovacuometer (Wika brand), dimensioned in cmH2O, with operating range ± 300 cmH2O, previously calibrated and equipped with pressure wall. Each operation will be repeated at least 5 and not more than 8 times, with the highest value being accepted, provided that the values do not exceed the value immediately below 10.

Fraction of expired Nitric Oxide:

Expiring Nitric Oxide Fraction (FENO)

The hay will be measured following the ATS criteria on the Mino NIOX ® (Aerocrine) equipment. Hay reading was performed on the reader, in parts per billion (ppb). To prevent air contamination of the sinus cavity, the procedure will be performed with nose clip.

Incremental Test:

Peripheral muscle strength will be performed by the 1RM test to determine the maximum training load. The incremental test will be conducted from upper limbs consisting of raising dumbbells diagonally, while for determination of lower limb load, bending and extension movements in Legpress. Before starting to test the children should be performed 5 to 10 repetitions, without load, to learn the movement properly and warm the muscles involved. The initial load used should be 0.5 kg and be progressively increased (0.5 kg) until the child reaches the maximum tolerated load, performing the full range of motion.

Treadmill Treadmill (Bruce Protocol):

The stress test, which provides information on exercise capacity and facilitates access to pathophysiological characteristics, drug efficacy and potential risk of disease, is best suited for children, physiologically has poorly developed knee extensors. And, for this reason, the ergometric test is preferred to the cycloergometer in young children (children from 4 to 6 years). The protocol used was that of Bruce who, although it was developed for adults, has been widely applied in children, from 4 years of age.

This protocol has been used to provide information on exercise capacity, pathophysiological characteristics during the fight, drug efficacy and potential risk of disease. The protocol will be discontinued only when the child reports fatigue or reaches the maximum heart rate around 195 to 205bpm. Throughout the test, blood pressure (BP) and peripheral oxygen saturation (SpO2) will be measured and an EKG will be done. The Borg scale will be used to quantify a sensation of shortness of breath during exertion and at rest.

Randomization:

Eligible children will be randomized into two different groups, one with video game training (VG) and the other associated with video game training for strength and resistance to upper limbs and lower limbs. (VGR). The allocation will be done through opaque, sealed and numbered envelopes. Two envelopes will be prepared for each participant. An envelope chosen by the patient to complete the revisions. The evaluation process will be conducted by a blind randomization and blind investigator who did not participate in the Protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged between 05 and 11 years
2. Both sexes
3. Diagnosis of asthma, according to the criteria of th e Global Initiative for Asthma (GINA)
4. Not be included in any program of regular physical activity
5. Not receiving Theophylline or aminophylline and oral steroid in the past 30 days
6. Not having presented with respiratory infection in the last 2 months
7. Have signed the term of free and clear in.

Exclusion Criteria:

1. Inability to understand or perform any one of the tests, due to physical and cognitive limitations
2. Intolerance the proposed activities
3. Be in in the presence of some infectious process with feverish and low adherence to the proposed Protocol

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Measurement of the Fraction of exhaled nitric oxide (FENO) | Change of Fraction of exhaled nitric oxide in 8 weeks at physical activity
  The fraction of exhaled nitric oxide (FENO) has been a feature used to complement the diagnosis of asthma in children and adults, in children are considered within normal values values up to 20 parts per billion (ppb). Patients with respiratory symptoms associated with FENO of 20ppb, which suggests the inflammation of the airways, may represent greater succession of seizures and non-control of the disease.
  The Fraction of exhaled nitric oxide will be measured by following the criteria of ATS, in the Mino NIOX ® equipment (Aerocrine).
  The evaluation of this variable will be performed prior to the therapeutic intervention and after 8 weeks in order to observe the level of airway inflammation after physical activity.
  An evaluation of this variable after 8 weeks of intervention aims to observe the level of inflammation of the airway and a physical activity.

SECONDARY OUTCOMES:
Measuring energy expenditure | Change in ability to exercise 8 weeks of physical activity
  Stress test (ET) is a diagnostic method with numerous indications in children and adolescents (age ≤ 19 years). This is considered the gold standard for determining exercise intolerance.
  The protocol chosen for this project is the Buce protocol. This protocol lasts 8 to 12 minutes, with small and constant increases in velocity and inclination, individualized for sex and age of the patient, based on the maximum expected oxygen consumption (VO2max), which can be estimated by the American College of Sports Medicine Formulas (ACSM) or the Veterans Specific-Activity Questionnaire (VSAQ).
  This test will be performed before and after a therapeutic treatment in order to observe an improvement in tolerance in a physical activity comparing two different protocols of physical activity.

CONTACTS AND LOCATIONS:
Locations (1):
- laboratory of Functional Respiratory Assessment, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided